CLINICAL TRIAL: NCT02112370
Title: Phase 3 Study of Ropivacaine (With Epinephrine) in BABA Endoscopic and Robotic Thyroidectomy
Brief Title: Efficacy of Ropivacaine (With Epinephrine) in BABA Endoscopic and Robotic Thyroidectomy
Acronym: REBT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Kyu Eun Lee, Associate Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B-1403/242-006
Record Dates: First submitted 2014-04-07; First posted 2014-04-11 (Estimated); Results first posted 2017-08-04 (Actual); Last update posted 2017-08-04 (Actual); Status verified 2017-04

CONDITIONS: Thyroid Neoplasm; Goiter
Keywords: Ropivacaine; Epinephrine; Endoscopy; Robotics; Thyroidectomy
MeSH Terms: conditions — Thyroid Neoplasms; Goiter | interventions — Ropivacaine; Epinephrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): 100cc normal saline is injected into the subcutaneous layer for the initial flap dissection.
  Interventions: Other: Placebo
- Ropivacaine with epinephrine injection (Experimental): 1 mg/mL 1cc epinephrine is diluted in 100cc normal saline and then 7.5 mg/mL 30cc ropivacaine is diluted in the same normal saline. The mixture is injected into the subcutaneous layer for the initial flap dissection.
  Interventions: Drug: Ropivacaine with epinephrine injection

INTERVENTIONS:
Drug: Ropivacaine with epinephrine injection — 1 mg/mL 1cc epinephrine is diluted in 100cc normal saline and then 7.5 mg/mL 30cc ropivacaine is diluted in the same normal saline. The mixture is injected into the subcutaneous layer for the initial flap dissection for the experiment group.
  Other Names: Hanlim ropiva injection 7.5 mg/mL (20cc); Insurance code: A37804211; Jeil epinephrine injection 1 mg/mL (1cc); Insurance code: A04900341
  Arms: Ropivacaine with epinephrine injection
Other: Placebo — 100cc normal saline is injected into the subcutaneous layer for the initial flap dissection for the placebo group.
  Other Names: CJ 0.9% Normal Saline injection 100cc; Insurance code: A11601752
  Arms: Placebo

SUMMARY:
To assess the pain relief and the hemodynamic stability of ropivacaine with epinephrine in BABA endoscopic and robotic thyroidectomy.

DETAILED DESCRIPTION:
Diluted ropivacaine with epinephrine is injected into the subcutaneous space to relieve pain and reduce bleeding during procedures. The synergistic effect of ropivacaine with epinephrine can contribute to patients' welfare, such as relieving pain and structuring the hemodynamic stability.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of thyroid neoplasm or benign goiter
* Scheduled for BABA endoscopic or robotic thyroidectomy

Exclusion Criteria:

* Completion thyroidectomy
* Modified radical neck dissection
* Allergy history
* Stroke history
* Uncontrolled hypertension
* Uncontrolled diabetes
* Coagulopathy
* Severe cardiovascular disease
* Severe pulmonary disease
* Chronic kidney disease
* Pregnant

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2014-05; Primary Completion 2016-05 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kyu Eun Lee, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (2):
- South Korea (2):
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Seoul National University Hospital, Seoul

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hristovska AM, Kristensen BB, Rasmussen MA, Rasmussen YH, Elving LB, Nielsen CV, Kehlet H. Effect of systematic local infiltration analgesia on postoperative pain in vaginal hysterectomy: a randomized, placebo-controlled trial. Acta Obstet Gynecol Scand. 2014 Mar;93(3):233-8. doi: 10.1111/aogs.12319. PMID 24576202
- [Background] Miratashi SA, Behdad S, Ayatollahi V, Ahmadi A. Hemodynamic effects of intraocular epinephrine during cataract surgery: a double blinded placebo controlled randomized clinical trial. Nepal J Ophthalmol. 2012 Jul-Dec;4(2):288-94. doi: 10.3126/nepjoph.v4i2.6546. PMID 22864036
- [Background] Kim SJ, Lee KE, Myong JP, Koo do H, Lee J, Youn YK. Prospective study of sensation in anterior chest areas before and after a bilateral axillo-breast approach for endoscopic/robotic thyroid surgery. World J Surg. 2013 May;37(5):1147-53. doi: 10.1007/s00268-013-1934-8. PMID 23397168
- [Background] Lee KE, Choi JY, Youn YK. Bilateral axillo-breast approach robotic thyroidectomy. Surg Laparosc Endosc Percutan Tech. 2011 Aug;21(4):230-6. doi: 10.1097/SLE.0b013e31822d0455. PMID 21857470
- [Background] Choe JH, Kim SW, Chung KW, Park KS, Han W, Noh DY, Oh SK, Youn YK. Endoscopic thyroidectomy using a new bilateral axillo-breast approach. World J Surg. 2007 Mar;31(3):601-6. doi: 10.1007/s00268-006-0481-y. PMID 17308853
- [Background] Choi JY, Lee KE, Chung KW, Kim SW, Choe JH, Koo do H, Kim SJ, Lee J, Chung YS, Oh SK, Youn YK. Endoscopic thyroidectomy via bilateral axillo-breast approach (BABA): review of 512 cases in a single institute. Surg Endosc. 2012 Apr;26(4):948-55. doi: 10.1007/s00464-011-1973-x. Epub 2011 Nov 4. PMID 22052422
- [Background] Kwon H, Koo do H, Choi JY, Kim E, Lee KE, Youn YK. Bilateral axillo-breast approach robotic thyroidectomy for Graves' disease: an initial experience in a single institute. World J Surg. 2013 Jul;37(7):1576-81. doi: 10.1007/s00268-013-2027-4. PMID 23558759
- [Background] Lee KE, Kim E, Koo do H, Choi JY, Kim KH, Youn YK. Robotic thyroidectomy by bilateral axillo-breast approach: review of 1,026 cases and surgical completeness. Surg Endosc. 2013 Aug;27(8):2955-62. doi: 10.1007/s00464-013-2863-1. Epub 2013 Feb 23. PMID 23436099
- [Background] Lee KE, Koo do H, Im HJ, Park SK, Choi JY, Paeng JC, Chung JK, Oh SK, Youn YK. Surgical completeness of bilateral axillo-breast approach robotic thyroidectomy: comparison with conventional open thyroidectomy after propensity score matching. Surgery. 2011 Dec;150(6):1266-74. doi: 10.1016/j.surg.2011.09.015. PMID 22136850
- [Background] Lee KE, Rao J, Youn YK. Endoscopic thyroidectomy with the da Vinci robot system using the bilateral axillary breast approach (BABA) technique: our initial experience. Surg Laparosc Endosc Percutan Tech. 2009 Jun;19(3):e71-5. doi: 10.1097/SLE.0b013e3181a4ccae. PMID 19542833
- [Derived] Lee JH, Suh YJ, Song RY, Yi JW, Yu HW, Kwon H, Choi JY, Lee KE. Preoperative flap-site injection with ropivacaine and epinephrine in BABA robotic and endoscopic thyroidectomy safely reduces postoperative pain: A CONSORT-compliant double-blinded randomized controlled study (PAIN-BREKOR trial). Medicine (Baltimore). 2017 Jun;96(22):e6896. doi: 10.1097/MD.0000000000006896. PMID 28562541
- See also: Pharmacology of regional anaesthesia — http://www.frca.co.uk/article.aspx?articleid=100816

RESULTS

PARTICIPANT FLOW:
Groups:
- Normal Saline Injection: 100cc normal saline is injected into the subcutaneous layer for the initial flap dissection.
  Placebo: 100cc normal saline is injected into the subcutaneous layer for the initial flap dissection.
- Ropivacaine With Epinephrine Injection: 1 mg/mL 1cc epinephrine is diluted in 100cc normal saline and then 7.5 mg/mL 30cc ropivacaine is diluted in the same normal saline. The mixture is injected into the subcutaneous layer for the initial flap dissection.
  Ropivacaine with epinephrine injection: 1 mg/mL 1cc epinephrine is diluted in 100cc normal saline and then 7.5 mg/mL 30cc ropivacaine is diluted in the same normal saline. The mixture is injected into the subcutaneous layer for the initial flap dissection.
Period: Overall Study
Arm/Group | Normal Saline Injection | Ropivacaine With Epinephrine Injection
Started | 74 | 74
Completed | 74 | 74
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All patients referred for BABA robotic or endoscopic thyroidectomy at Seoul National University Bundang Hospital
Groups:
- Total: Total of all reporting groups
Arm/Group | Normal Saline Injection | Ropivacaine With Epinephrine Injection | Total
Number analyzed (Participants) | 74 | 74 | 148
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.0 (9.3) | 35.5 (8.8) | 36.1 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69 | 66 | 135
  Male | 5 | 8 | 13
Preoperative thyroid function test (T3, ng/dL) [Mean (Standard Deviation); unit: ng/dL] | 121.8 (15.0) | 123.3 (25.1) | 122.5 (20.6)
Preoperative thyroid function test (free T4, ng/dL) [Mean (Standard Deviation); unit: ng/dL] | 1.2 (0.3) | 1.2 (0.4) | 1.2 (0.4)
Preoperative thyroid function test (TSH, uIU/mL) [Mean (Standard Deviation); unit: uIU/mL] | 1.8 (1.0) | 2.2 (1.7) | 2.0 (1.4)
Method of operation (robotic/endoscopic) [Number; unit: participants]
  Robotic | 53 | 55 | 108
  Endoscopic | 21 | 19 | 40
Extent of operation (Right/Left/Total) [Number; unit: participants]
  Right | 26 | 29 | 55
  Left | 28 | 24 | 52
  Total | 20 | 21 | 41

OUTCOME MEASURES:

1. Primary Outcome: NRS Pain Scores for the First 12 Hours
Description: The numerical rating scale is utilized to assess the postoperative pain change for the first 12 hours according to location.
  Range: 0(minimal pain, better outcome) ~ 10(maximum pain, worse outcome)
  Unlike the general NRS pain score as reported in the "post-operative 48 hour" result which deals with post-operative discomfort in general, this outcome measures the pain score of the specific location in which flap dissection had taken place.
Time Frame: Postoperative 12 hours
Measure: Mean (Standard Deviation); unit: points
Arm/Group | Normal Saline Injection | Ropivacaine With Epinephrine Injection
Number analyzed (Participants) | 74 | 74
points
  Swallowing difficulty | 4.93 (1.79) | 4.12 (1.87)
  Anterior neck pain | 4.50 (2.10) | 3.69 (1.94)
  Right chest pain | 3.99 (2.27) | 3.16 (1.96)
  Left chest pain | 3.74 (1.94) | 4.51 (2.45)
  Back pain | 0.65 (1.50) | 0.28 (1.05)
  Posterior neck pain | 1.47 (2.07) | 1.65 (2.40)
Statistical Analysis 1: Comparison: Normal Saline Injection vs Ropivacaine With Epinephrine Injection; Swallowing difficulty; Test type: Superiority or Other; p = 0.008, t-test, 2 sided — threshold p value for significance < 0.05
Statistical Analysis 2: Comparison: Normal Saline Injection vs Ropivacaine With Epinephrine Injection; Anterior neck pain; Test type: Superiority or Other; p = 0.016, t-test, 2 sided — threshold p value for significance < 0.05
Statistical Analysis 3: Comparison: Normal Saline Injection vs Ropivacaine With Epinephrine Injection; Right chest pain; Test type: Superiority or Other; p = 0.019, t-test, 2 sided — threshold p value for significance < 0.05
Statistical Analysis 4: Comparison: Normal Saline Injection vs Ropivacaine With Epinephrine Injection; Left chest pain; Test type: Superiority or Other; p = 0.035, t-test, 2 sided — threshold p value for significance < 0.05
Statistical Analysis 5: Comparison: Normal Saline Injection vs Ropivacaine With Epinephrine Injection; Back pain; Test type: Superiority or Other; p = 0.089, t-test, 2 sided — threshold p value for significance < 0.05
Statistical Analysis 6: Comparison: Normal Saline Injection vs Ropivacaine With Epinephrine Injection; Posterior neck pain; Test type: Superiority or Other; p = 0.634, t-test, 2 sided — threshold p value for significance < 0.05

2. Secondary Outcome: Maximum of Measured Systolic Blood Pressures
Description: The maximal systolic blood pressure is monitored during surgery.
Time Frame: participants were followed for the duration of the operation, an average of approximately 2.5 hours
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Normal Saline Injection | Ropivacaine With Epinephrine Injection
Number analyzed (Participants) | 74 | 74
mmHg | 142 (16.5) | 145 (18.9)

3. Secondary Outcome: Maximum of Measured Diastolic Blood Pressures
Description: The maximal diastolic blood pressure is monitored during surgery.
Time Frame: participants were followed for the duration of the operation, an average of approximately 2.5 hours
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Normal Saline Injection | Ropivacaine With Epinephrine Injection
Number analyzed (Participants) | 74 | 74
mmHg | 91 (14.9) | 86 (19.2)

4. Secondary Outcome: Maximum of Measured Heart Rates
Description: The maximal heart rate is monitored during surgery.
Time Frame: participants were followed for the duration of the operation, an average of approximately 2.5 hours
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Normal Saline Injection | Ropivacaine With Epinephrine Injection
Number analyzed (Participants) | 74 | 74
beats per minute | 88 (16.1) | 99 (13.3)

5. Secondary Outcome: Blood Loss Amount
Description: The blood loss amount is estimated at the end of surgery.
Time Frame: participants were followed for the duration of the operation, an average of approximately 2.5 hours
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Normal Saline Injection | Ropivacaine With Epinephrine Injection
Number analyzed (Participants) | 74 | 74
ml | 30 (58.2) | 18 (40.5)

6. Secondary Outcome: Operation Time
Description: The amount of time taken from start to the end of surgery
Time Frame: participants were followed for the duration of the operation, an average of approximately 2.5 hours
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Normal Saline Injection | Ropivacaine With Epinephrine Injection
Number analyzed (Participants) | 74 | 74
minutes | 163.6 (54.1) | 155.3 (46.8)

7. Secondary Outcome: NRS Change
Description: Change in NRS score a with time The numerical rating scale is utilized to assess the postoperative pain change for the first 12 hours according to location.
  Range: 0(minimal pain, better outcome) ~ 10(maximum pain, worse outcome)
Time Frame: 0, 1, 2, 4, 6, 9, 12, 24, and 48 hours post operation
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Normal Saline Injection | Ropivacaine With Epinephrine Injection
Number analyzed (Participants) | 74 | 74
scores on a scale
  0 hour | 5.73 (2.02) | 5.68 (2.13)
  1 hour | 5.05 (1.95) | 4.7 (1.59)
  2 hour | 4.55 (1.80) | 4.11 (1.56)
  4 hour | 3.55 (1.27) | 3.34 (1.19)
  6 hour | 3.39 (1.29) | 3.28 (1.22)
  9 hour | 3.28 (1.34) | 3.14 (1.38)
  12 hour | 3.19 (1.37) | 3.18 (1.23)
  24 hour | 2.93 (1.09) | 2.95 (1.05)
  48 hour | 2.27 (0.94) | 2.08 (0.90)

8. Secondary Outcome: Pain Killer Dose
Description: Change in pain killer usage with time
Time Frame: 0, 1, 2, 4, 6, 9, 12, 24, and 48 hours post operation
Measure: Mean (Standard Deviation); unit: vials (15mg ketorolac per vial)
Arm/Group | Normal Saline Injection | Ropivacaine With Epinephrine Injection
Number analyzed (Participants) | 74 | 74
vials (15mg ketorolac per vial)
  0 hour | 1 (0.72) | 0.84 (0.60)
  1 hour | 0.35 (0.51) | 0.31 (0.47)
  2 hour | 0.31 (0.49) | 0.26 (0.44)
  4 hour | 0.07 (0.25) | 0.11 (0.31)
  6 hour | 0.18 (0.38) | 0.15 (0.36)
  9 hour | 0.14 (0.34) | 0.12 (0.33)
  12 hour | 0.18 (0.42) | 0.19 (0.43)
  24 hour | 0.20 (0.44) | 0.16 (0.41)
  48 hour | 0.01 (0.11) | 0.07 (0.15)

ADVERSE EVENTS:
Arm/Group | Normal Saline Injection | Ropivacaine With Epinephrine Injection
Serious Adverse Events (participants affected / at risk) | 0/74 | 0/74
Other Adverse Events (participants affected / at risk) | 0/74 | 0/74

LIMITATIONS AND CAVEATS:
1. Single-institution study
2. We did not directly examine the vasoconstrictive properties of epinephrine in helping reduce bleeding.
3. Issue regarding importance of statistical vs. clinical significance of the pain score remains to be addressed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No